CLINICAL TRIAL: NCT06824857
Title: Effect of Postoperative Abdominal Massage on Bowel Movements in Patients With Subarachnoid Hemorrhage
Brief Title: Effect of Abdominal Massage on Bowel Movements in Patients With Subarachnoid Hemorrhage
Acronym: Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zühal Erdoğan, RN, PhD, Assistant Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024 - 306
Record Dates: First submitted 2024-10-11; First posted 2025-02-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Subarachnoid Haemorrhage (SAH)
Keywords: subarachnoid hemorrhage; Abdominal massage; bowel movements; nursing
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Massage Application Group (Experimental): After explaining the purpose of the study to the relatives of patients in the abdominal massage group, the "Introductory Characteristics Form" will be filled out. Abdominal massage will be performed according to the Checklist at the 6th hour after surgery and at the same times in the morning and evening for the first 3 days post-surgery. Before and 15 minutes after the abdominal massage application, bowel sounds will be auscultated, abdominal circumference will be measured with a measuring tape, and abdominal tension will be observed and recorded in the patient follow-up form.
  Interventions: Other: Abdominal Massage Application
- Control Group (No Intervention): After explaining the purpose of the study to the relatives of patients in the control group, the "Introductory Characteristics Form" will be filled out. At the same times as the experimental group, bowel sounds will be auscultated in the control group without any intervention, abdominal circumference will be measured with a measuring tape, and abdominal tension will be observed

INTERVENTIONS:
Other: Abdominal Massage Application — As part of the abdominal massage application, patient follow-up forms and checklists were prepared. Before starting the study, the abdominal massage practitioner participated in a certification program on this topic and received a competency certificate. Patients will be followed up for the first 3 days postoperatively using the prepared patient follow-up forms. Abdominal massage will be applied to each patient for 15 minutes according to a certain standard as stated in the literature
  Arms: Abdominal Massage Application Group

SUMMARY:
The study will be conducted as a randomized controlled trial to determine the effect of postoperative abdominal massage on bowel movements in patients who underwent surgery after subarachnoid hemorrhage and are hospitalized in the neurosurgery intensive care unit.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled trial to determine the effect of postoperative abdominal massage on bowel movements in patients who underwent surgery after subarachnoid hemorrhage and are hospitalized in the neurosurgery intensive care unit. The sample of the study will consist of a total of 64 patients, 32 in the experimental group and 32 in the control group, hospitalized in the tertiary neurosurgery intensive care unit. Data collection tools are the "Descriptive Characteristics Form" and the "Patient Follow-up Form".The statistician will determine whether the patients who meet the sampling criteria will be assigned to the experimental or control group through randomization. The stratified randomization method will be used in the study. In this context, patients who meet the inclusion criteria from the start date of the study in the Neurosurgery Intensive Care Unit will be randomized by assigning them to the control group and abdominal massage groups, respectively. Patients will be assigned to the control and abdominal massage groups in this order until the sample size is reached. The CONSORT diagram will be used in the randomization of patients.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older

  * Underwent neurovascular surgery
  * Received general anesthesia
  * Have no wounds, surgical intervention, or radiotherapy in the abdominal region
  * Have no bowel obstruction, irritable bowel syndrome, inflammatory bowel disease, abdominal herniation, or bowel cancer
  * Began oral feeding at the 6th hour post-surgery
  * Stayed in the intensive care unit for 3 or more days
  * Have a Glasgow Coma Scale (GCS) score of 9 or above
  * Have no signs of acute abdomen
  * Have no intra-abdominal infection
  * No mechanical ventilation
  * Mobilezed in the preoperative period
  * Unable to mobilize after surgery
  * Evaluated by the intensive care physician with no contraindications for abdominal massage
  * Have a first-degree relative who has given consent

Exclusion Criteria:

* Patients with the following conditions will be excluded from the sample:

  * Those with chronic constipation, fecal incontinence, or diarrhea
  * Those fed with a fiber-enriched nutritional solution (e.g., Nutrison Protein Plus Multifibre®, Fresubin Original Fibre®, Isosource Fiber®, Jevity Plus®)
  * Those fed via nasogastric enteral tube
  * Those receiving parenteral nutrition
  * Patients with a BMI > 40 (morbid obesity)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Time To Defecate | From the 6th hour after surgery until the end of the 3rd day after surgery
  Time of first defecation
Bowel Sounds | From the 6th hour after surgery until the end of the 3rd day after surgery
  Frequency of bowel sounds heard per minute
Abdominal Distension | From the 6th hour after surgery until the end of the 3rd day after surgery
  To be assessed by measuring the abdominal circumference with a tape measure

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Nursing, Gazi University, Ankara
  - Gazi University, Ankara

IPD SHARING:
Plan to Share IPD: No